CLINICAL TRIAL: NCT04365413
Title: A Feasibility Study for the Use of Multispectral Optoacoustic Tomography in the Detection of Solid Tumors and Lymph Nodes (MSOT)
Brief Title: A Feasibility Study for the Use of Multispectral Optoacoustic Tomography in the Detection of Tumors
Acronym: OU-SCC-MSOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OU-SCC-MSOT
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor
Keywords: Imaging device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Imaging of Tumor or Lymph node (Experimental): Tumors and/or lymph nodes of patients scheduled for standard of care surgery will be imaged using the MSOT device before and after surgery.
  The temperature of their skin prior to and after MSOT imaging will also be measured.
  Interventions: Device: MSOT Device; Procedure: Temperature Measurement

INTERVENTIONS:
Device: MSOT Device — The MSOT Device will be used to take images of the tumor and/or lymph nodes of patients with solid tumors before and after surgery to measure the margins of the tumor and/or positive lymph node.
Procedure: Temperature Measurement — The temperature of the skin will be measured prior to and after MSOT imaging.

SUMMARY:
The purpose of this study is to evaluate the safety and potential of a new experimental imaging instrument called multispectral optoacoustic tomography (MSOT) to detect tumors and lymph nodes with tumors.

DETAILED DESCRIPTION:
This study will involve patients that are scheduled for routine standard of care surgery. It is a single-arm study designed to provide safety information regarding the use of the Acuity MSOT device in the clinical setting, and the ability of MSOT imaging data to correlate with clinical findings identified via pathology.

The device will be used to obtain images of the tumor or lymph node margins for investigational use only to compare to clinical pathology and patient's medical record. All images will be obtained pre- and post-surgery in a closed surgical patient. The temperature of the patient's skin will also be measured prior to and after MSOT imaging. MSOT imaging will be for research only and no treatment decisions will be based on the MSOT images obtained.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an identified solid tumor, i.e. breast (Stage I-IV), melanoma (Stage I-IV), HNSCC (Stage I-III), pancreatic (Stage I-III), ovarian (Stage I-IV) that is scheduled for surgical removal of the tumor and completed standard imaging prior to surgery
* Have acceptable hematologic status [total hemoglobin (tHb) ≥ 10 mg/dL]
* Patients ≥ 18 yrs of age
* Patient provided a signed and dated informed consent
* Willing to comply with study procedures and be available for the duration of the study
* Ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

* Patients with central nervous system tumors
* Patients with a tattoo over the surgical site
* Pregnant women
* Women who are breastfeeding
* Systemic or local infection
* Any systemic anomaly during the pre-op assessment preventing patient participation in the study
* Any febrile illness that precludes or delays participation preoperatively
* Anything that would put the participant at increased risk or preclude compliance with the study
* Patients with Stage IV pancreatic cancer, Stage IV HNSCC are not surgical candidates and therefore excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lacey McNally, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled on this study at the University of Oklahoma Stephenson Cancer Center between July 2020 and July 2021. The first participant was enrolled on July 22th, 2020 and the last participant was enrolled on July 12th, 2021.
Pre-assignment Details: Of the 54 enrolled participants, 49 participants met the inclusion criteria, and 5 were designated as screen fails. Of the 49 participants, 45 were assigned to be scanned by the MSOT device and had skin temperature measurements taken, and 4 did not continue on the study.
Groups:
- Imaging of Tumor or Lymph Node Using MSOT and Temperature Measurement: The MSOT Device was used to take images of the tumor and/or lymph nodes of patients with solid tumors before and after surgery to measure the margins of the tumor and/or positive lymph node.
  The temperature of the skin was measured prior to and after MSOT imaging.
Period: Overall Study
Arm/Group | Imaging of Tumor or Lymph Node Using MSOT and Temperature Measurement
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Any participant who met inclusion criteria.
Groups:
- Imaging of Tumor or Lymph Node: Tumors and/or lymph nodes of patients scheduled for standard of care surgery will be imaged using the MSOT device before and after surgery.
  The temperature of their skin prior to and after MSOT imaging will also be measured.
  MSOT Device: The MSOT Device will be used to take images of the tumor and/or lymph nodes of patients with solid tumors before and after surgery to measure the margins of the tumor and/or positive lymph node.
  Temperature Measurement: The temperature of the skin will be measured prior to and after MSOT imaging.
Arm/Group | Imaging of Tumor or Lymph Node
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.59 (11.848)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 37
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Weight for two patients was not collected.
  kg/m^2
    number analyzed (Participants) | 47
    (all) | 30.15 (7.485)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Due to MSOT Imaging
Description: Adverse events as characterized by CTCAE v5.0 in patients that may result from MSOT imaging (≥44 degrees Celsius).
  Measurement of skin temperature pre- and post-MSOT imaging (2 measurements total) with a touch thermometer as part of the safety evaluation of the MSOT device. The thermometer will be placed onto the skin until a temperature appears, about 1 minute, and the temperature will be recorded.
Time Frame: 1-2 minutes
Population: Patients who completed pre and post MSOT imaging temperature readings.
Measure: Count of Participants; unit: Participants
Arm/Group | Imaging of Tumor or Lymph Node
Number analyzed (Participants) | 45
Participants | 0

2. Primary Outcome: Evaluate Skin Temperature Pre and Post Imaging (Pre- and Post- Surgery)
Description: Percent of patients who experienced skin temperature readings >44 degrees Celsius.
Time Frame: 1-2 minutes after imaging
Measure: Number; unit: Percent of patients
Arm/Group | Imaging of Tumor or Lymph Node
Number analyzed (Participants) | 45
Percent of patients | 0

3. Secondary Outcome: Tumor Positivity Based on Detection of Oxy-hemoglobin Using MSOT Device.
Description: MSOT device can identify and differentiate between tumor tissue and surrounding tissue due to detection of different oxygenation states of hemoglobin, with the idea that tumors have differential tissue oxygenation levels compared to non-tumor (control) values. Tumor positivity will be determined based on comparison of oxy-hemoglobin levels using MSOT localization from the same size polygon region of interest (ROI) analysis of the tumor tissue and a sample of non-cancer tissue from the same patient. Increased intensity of signal (output obtained in MSOT Arbitrary Units (MSOT A.U.)) indicates higher levels of oxy-hemoglobin which correlates with tumor tissue as confirmed by comparison with pathology reports. Paired t-tests will be performed and median difference and IQR reported.
Time Frame: 6 months
Population: Patients who underwent MSOT scanning who had usable data (no machine errors)
Measure: Median (Inter-Quartile Range); unit: MSOT A. U.
Arm/Group | Imaging of Tumor or Lymph Node
Number analyzed (Participants) | 43
MSOT A. U. | 0.0687 [0.0407 to 0.1019]
Statistical Analysis 1: Comparison: Imaging of Tumor or Lymph Node; Test type: Other; p < 0.0001, Paired t-test; Median Difference (Final Values) = 0.069

4. Secondary Outcome: Tumor Positivity Based on Detection of Deoxy-hemoglobin Using MSOT
Description: MSOT device can identify and differentiate between tumor tissue and surrounding tissue due to detection of different oxygenation states of hemoglobin, with the idea that tumors have differential tissue oxygenation levels compared to non-tumor (control) values. Tumor positivity will be determined based on comparison of deoxy-hemoglobin levels using MSOT localization from the same size polygon region of interest (ROI) analysis of the tumor tissue and a sample of non-cancer tissue from the same patient. Increased intensity of signal (output obtained in MSOT Arbitrary Units (MSOT A.U.)) indicates higher levels of deoxy-hemoglobin which correlates with tumor tissue as confirmed by comparison with pathology reports. Paired t-tests will be performed and median difference and IQR is reported.
Time Frame: 6 months
Population: Patients who underwent MSOT scanning who had usable data (no machine errors)
Measure: Median (Inter-Quartile Range); unit: MSOT A. U.
Arm/Group | Imaging of Tumor or Lymph Node
Number analyzed (Participants) | 43
MSOT A. U. | 0.0420 [0.0293 to 0.0845]
Statistical Analysis 1: Comparison: Imaging of Tumor or Lymph Node; Test type: Other; p < 0.0001, Paired t-test; Median Difference (Final Values) = 0.042

5. Secondary Outcome: Tumor Positivity From Pathology Reports Compared to MSOT Readings
Description: Tumor positivity will be compared (yes/no) from the standard pathology report with the MSOT readings. Percent of patients with matching readings will be calculated and reported.
Time Frame: 6 months
Population: Patients with pathology reports and viable MSOT readings
Measure: Number; unit: percent of patients
Arm/Group | Imaging of Tumor or Lymph Node
Number analyzed (Participants) | 43
percent of patients | 100

ADVERSE EVENTS:
Time Frame: 31 days
Description: A slight, reversible reddening and temperature increase of sensitive skin. All adverse events and expected treatment effects, including mild events, will be monitored throughout the study until discharge.
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting.
Arm/Group | Imaging of Tumor or Lymph Node
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT04365413/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT04365413/SAP_001.pdf
  • Informed Consent Form (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT04365413/ICF_002.pdf